CLINICAL TRIAL: NCT04152057
Title: A Single-arm, Exploratory Clinical Study of Pyrotinib Maleate Tablets Combined With Albumin Paclitaxel and Trastuzumab for Her2-positive Early or Locally Advanced Breast Cancer and Its Biomarkers
Brief Title: Pyrotinib Maleate Tablets Combined With Albumin Paclitaxel and Trastuzumab for Her2-positive Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shuangyue Liu, Assisting staff, West China Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLTN-NeoBC1115
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer; HER2 Positive; Combination Chemotherapy
Keywords: Pyrotinib Maleate Tablets; Trastuzumab; Albumin Paclitaxel; Early or Locally Advanced; neoadjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib Combined With Albumin Paclitaxel and Trastuzumab (Experimental): Preoperative
  -Drug: Pyrotinib Maleate Tablets combined with Albumin Paclitaxel and Trastuzumab.
  Surgery:Subjects should be evaluated by tumor-enhanced MRI combined with mammary gland ultrasound during the preoperative neoadjuvant administration, and evaluated every 2 cycles. The subjects who were evaluated for CR and PR for the first time should be confirmed after at least 4 weeks. The confirmed tumor assessment cannot change the previously fixed examination time point.
  Postoperative
  * Drug: Epirubicin hydrochloride combined with Cyclophosphamide
  * At the same time, according to the recommendation of the clinician, choose whether to accept the same anti-HER2 treatment plan before surgery. For patients with tumors positive for estrogen receptor (ER) and/or progesterone receptor (PR), endocrine therapy should be given at the end of adjuvant chemotherapy, and if there is clinical indication at the end of adjuvant chemotherapy, radiotherapy should be given.
  Interventions: Drug: Pyrotinib Maleate Tablets; Drug: Albumin Paclitaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: Pyrotinib Maleate Tablets — 400mg/d,po qd,q3w, 4 cycles
  Other Names: Malaisuan Biluotini Pian; Ai Rui Ni
Drug: Albumin Paclitaxel — 125mg/m2,ivggt,d1,q3w,4 cycles.
  Other Names: Ai Yue
Drug: Trastuzumab — The first week load dose 4mg / kg, followed by 2mg / kg per week, d1,ivggt,q3w,4 cycles.
  Other Names: Qutuozhu DanKang; Herceptin

SUMMARY:
This study was designed to evaluate the efficacy and safety of pyrotinib combined with albumin paclitaxel and trastuzumab in the treatment of Her2-positive early or locally advanced breast cancer, and to explore RCB scores and TILs expression and other related molecular markers for pyrrole the efficacy of the treatment with pyrotinib.

DETAILED DESCRIPTION:
At present, the treatment mode of breast cancer has gradually turned to the individualized comprehensive treatment mode combining systemic therapy and local therapy, and neoadjuvant therapy is widely used. Albumin-bound paclitaxel alters the excipients, reduces adverse reactions and greatly enhances efficacy, facilitating clinical applications. Studies have shown that in the use of neoadjuvant chemotherapy, drugs containing purple shirts and anthracyclines will be the drug of choice. The HER2/erbB2 molecule is an independent prognostic factor for breast cancer. About 20%-30% of adenocarcinoma patients have amplification/overexpression of HER2 gene. These patients are insensitive to conventional therapy and are more prone to recurrence and metastasis. Shorter survival and poorer prognosis. Current drugs targeting HER2 targets mainly include macromolecular monoclonal antibodies and their conjugates and small molecule tyrosine kinase inhibitors. Pyrotinib is an irreversible inhibitor of small targets (EGFR and HER2). Compared with trastuzumab, it has different sites of action, which may lead to synergy in the treatment of human Her2-positive breast cancer.

The excellent clinical efficacy of dual-targeted neoadjuvant therapy for Her2 positive breast cancer, the anti-tumor effect and good tolerance of pyrotinib, we intend to develop a pyrotinib combined with albumin paclitaxel and trastuzumab one-arm exploratory clinical study of neoadjuvant therapy for Her2-positive early or locally advanced breast cancer with the aim of assessing efficacy and safety, and exploring the efficacy of tumor-associated molecular markers such as RCB scores and TILs expression for pyrotinib treatment predicting effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, and ≤ 70 years old .
* ECOG full body status 0-1 .
* According to the RECIST 1.1 standard, at least one measurable lesion exists.
* The pathological examination confirmed the positive expression of HER2, the clinical stage was stage II-III [cT2 and any N, cT3 and any N; cT4 and any N, according to the American Joint Committee on Cancer (AJCC) criteria] breast cancer patients .

Note: HER2 expression positive refers to the pathological detection/review of primary or metastatic lesions performed by the pathology department of the Institute of Research and Development, at least once, at least 10% of tumor cells have immunohistochemical staining intensity of 3+ [staining intensity] Range 0 to 3] or positive by fluorescence in situ hybridization [FISH].

* The functional level of organs must meet the following requirements: ANC≥1.5×10E+9/L,PLT≥90×10E+9/L,Hb≥90 g/L,TBIL≤1.5×ULN,ALT 和 AST≤2×ULN,BUN 和 Cr≤ 1.5×ULN 且Creatinine clearance ≥50 mL/min（Cockcroft-Gault）.Echocardiography:LVEF≥50%,12-lead ECG:The QT interval (QTcF) corrected by the Fridericia method was < 450 ms for males and < 470 ms for females.
* Patients with known hormone receptor status .
* In patients with a negative serum pregnancy test, patients with fertility potential must agree to use an effective non-hormonal contraceptive method during treatment and at least 6 months after the last use of the test drug.
* Volunteered to join the study, signed informed consent, had good compliance and was willing to cooperate with follow-up.

Exclusion Criteria:

Not selected as a subject in any of the following circumstances

* Patients with inflammatory breast cancer .
* Patients with metastatic breast cancer (stage IV) .
* Unable to swallow, chronic diarrhea and intestinal obstruction, there are many factors affecting the administration and absorption of drugs .
* Patients who received radiotherapy, chemotherapy, surgery (large surgery for breast cancer) or molecular targeted therapy 4 weeks before randomization were randomized to receive endocrine therapy within 7 days prior to randomization.
* Participated in other drug clinical trials within 4 weeks before randomization .
* The body has previously used or is using HER2-targeted monoclonal antibodies or tyrosine kinase inhibitor (including Trastuzumab,Pertuzumab,Lapatinib,Linatinib and Pyrotinib).
* Has had other malignant tumors in the past 5 years, excluding cured cervical carcinoma in situ, cutaneous basal cell carcinoma or cutaneous squamous cell carcinoma.
* Also accept any other anti-tumor treatment .
* Known to have a history of allergies to the drug components of this regimen; history of immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency disease, or history of organ transplantation .
* Have had any heart disease, including: (1) angina; (2) drug-treated or clinically significant arrhythmia; (3) myocardial infarction; (4) heart failure; (5) any subject judged Other heart diseases that are not suitable for this trial, etc.
* Female patients in pregnancy or lactation, female patients with fertility and positive pregnancy test, or women of childbearing age who are unwilling to take effective contraceptive measures during the whole trial period.
* According to the investigator's judgment, there are serious concomitant diseases that are harmful to the patient's safety or affect the patient's completion of the study (including but not limited to severe hypertension, severe diabetes, active infection, etc. that the drug cannot control).
* Have a clear history of neurological or mental disorders, including epilepsy or dementia.
* Accompanying CYP3A4 inhibitor or inducer .
* The investigator believes that the patient is not eligible for any other study in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
pathologic Complete Response(pCR)（ypT0/is N0） | Postoperative evaluation after completion of neoadjuvant therapy (approximately 24 weeks) .
  Invasive tumor residuals in the breast and axillary lymph nodes without microscopic examination, ductal carcinoma in situ may exist.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to 2 years
  The proportion of patients with a best overall confirmed response of CR or PR in the whole body as assessed per RECIST 1.1 by the investigator.
Disease Control Rate (DCR) | up to 2 years
  The proportion of patients with a best overall response of CR, PR or SD in the whole body, as assessed per RECIST1.1 by the investigator.
Residual Cancer Burden (RCB) | up to 2 years
  The RCB category (RCB-0, RCB-I, RCB-II, or RCB-III) was defined according to the M.D. Anderson Cancer Center standard, and the RCB score was associated with the patient's prognosis.
Tumor Infiltrating Lymphocytes (TILS) | up to 2 years
  This outcome measure is designed to measure the amount of TILs in newly diagnosed luminal A and Triple Negative Breast Cancer (TNBC) tumors. The mean percent change in TILS in tumor tissue from initial core biopsy samples will be compared with pathology samples from definitive surgery after IORT between the two different breast cancer sub types.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Luo, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Chengdu, Sichuan, China, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhong X, He P, Chen J, Yan X, Wei B, Zhang Z, Bu H, Li J, Tian T, Lv Q, Wang X, Li H, Wang J, Huang J, Suo J, Liu X, Zheng H, Luo T. Neoadjuvant pyrotinib plus trastuzumab and nab-paclitaxel for HER2-positive early or locally advanced breast cancer: an exploratory phase II trial. Gland Surg. 2022 Jan;11(1):216-225. doi: 10.21037/gs-21-911. PMID 35242683